CLINICAL TRIAL: NCT00952315
Title: Randomized Controlled Trial Comparing Three Different Modalities of Newer Lithotrites For Intracorporeal Lithotripsy
Brief Title: Trial Comparing Three Different Devices for Kidney Stone Removal During Percutaneous Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana Kidney Stone Institute (Other)
Responsible Party: Principal Investigator, James Lingeman, James Lingeman, MD, Indiana Kidney Stone Institute
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 09-045
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Kidney Stones
Keywords: kidney stones; intracorporeal lithotriptors; kidney stone removal
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stonebreaker (Active Comparator): Stonebreaker will be used to break up the kidney stone. Duration will be timed and documented.
  Interventions: Device: Stonebreaker
- Lithoclast Select (Active Comparator): Lithoclast Select will be used to breakup and remove kidney stone. Duration will be timed and documented.
  Interventions: Device: Lithoclast Select
- Cyberwand (Active Comparator): The dual probe Cyberwand device will be used to fragment and remove the kidney stone. Duration will be timed and documented.
  Interventions: Device: Cyberwand

INTERVENTIONS:
Device: Cyberwand — Dual probe lithotrite Cyberwand will be used to remove kidney stone. Duration will be timed and documented.
  Arms: Cyberwand
Device: Stonebreaker — Stonebreaker will be used to break up the kidney stone. Duration will be timed and documented.
  Arms: Stonebreaker
Device: Lithoclast Select — Lithoclast Select will be used to break up and remove the kidney stone. Duration will be timed and documented
  Arms: Lithoclast Select

SUMMARY:
The investigators plan to compare three different devices that are used to break up large kidney stones during surgery for removal to see if one is faster or more efficient than the others.

DETAILED DESCRIPTION:
Large kidney stones can be removed by a surgical procedure where a small puncture is made through the back into the kidney (percutaneous nephrolithotomy or PNL) but the stones usually need to be broken into smaller pieces before they can be removed through the small surgical incision. There are a number of FDA approved devices commercially available used to break up the stones including pneumatic, ultrasonic, and a combination of the two. Each technology has advantages and disadvantages.

In the last few years there have been new, improved versions of these devices introduced. These improved versions have addressed previous issues of probes clogging or breaking and cumbersome handpiece design. These include the Cyberwand (Cybersonics, Erie, PA), a dual probe ultrasonic device, Swiss Lithoclast Select (EMS, Switzerland) combining the pneumatic and ultrasonic modalities, and a novel device by LMA (Gland, Switzerland) called the StoneBreakerTM, a portable pneumatic device powered by CO2 cartridges.

We propose to compare each of these devices in a randomized study to see if one is better than another at removing kidney stones quickly and efficiently.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo percutaneous nephrolithotomy for at least one kidney stone measuring 2 cm or greater
* Stone easily visible/measurable on plain abdominal imaging (KUB) or CT scan preoperatively
* Age 18 years or older
* Able to give informed consent

Exclusion Criteria:

* Size of single largest stone less than 2 cm
* Pregnancy
* Active urinary tract infection
* Extracorporeal shockwave lithotripsy within the last three months
* Complex stone anticipating multiple access sites
* Stones that are not clearly able to be measured on KUB or CT scan
* Inability to give informed consent
* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2009-08; Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Lingeman, MD, Principal Investigator — IU Health Physicians Urology
Locations (10):
- United States (8):
  - Mayo Clinic Scottsdale, Phoenix, Arizona
  - Northwestern University, Chicago, Illinois
  - IU Health Physicians Urology, Indianapolis, Indiana
  - Johns Hopkins, Baltimore, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Duke University, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Wisconsin, Madison, Wisconsin
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - The University of Western Ontario, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: International Kidney Stone Institute - Click here for more information about kidney stone disease — http://iksi.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand
Started | 90 | 90 | 90
Completed | 64 | 66 | 71
Not Completed | 26 | 24 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand | Total
Number analyzed (Participants) | 64 | 66 | 71 | 201
Age, Continuous [Mean (Full Range); unit: years] | 55.2 [22 to 80] | 58.1 [20 to 83] | 57.4 [24 to 89] | 57 [20 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 34 | 36 | 102
  Male | 32 | 32 | 35 | 99
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  North America | 64 | 66 | 71 | 201

OUTCOME MEASURES:

1. Primary Outcome: Stone Clearance Time in mm2/Min
Description: Clearance rate was calculated by dividing the surface area of the targeted stone (mm2) by the total clearance time (min)
Time Frame: collected intraoperatively from the time stone breakage begins to end of stone removal with a stone extraction basket
Measure: Mean (Standard Deviation); unit: mm^2/min
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand
Number analyzed (Participants) | 64 | 66 | 71
mm^2/min | 24.0 (13.9) | 28.9 (16.2) | 32.3 (23.4)

2. Secondary Outcome: Stone-free After First Procedure
Description: Number of participants deemed stone-free after initial stone-removal surgery
Time Frame: Post-operative Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand
Number analyzed (Participants) | 64 | 66 | 71
Participants | 33 | 43 | 39

3. Secondary Outcome: Secondary Procedure Required
Description: Number of participants who required a secondary kidney stone removal procedure
Time Frame: Within three days of initial procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand
Number analyzed (Participants) | 64 | 66 | 71
Participants | 15 | 16 | 24

4. Secondary Outcome: Ureteral Stent Placed
Description: Participants requiring a ureteral stent to be placed after initial stone removal procedure
Time Frame: Intra-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand
Number analyzed (Participants) | 64 | 66 | 71
Participants | 3 | 4 | 5

5. Secondary Outcome: Nephrostomy Tube Placed
Description: Participants requiring a nephrostomy tube to be placed at the end of the initial stone removal procedure
Time Frame: Intra-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand
Number analyzed (Participants) | 64 | 66 | 71
Participants | 55 | 59 | 63

6. Secondary Outcome: Use of Other Device
Description: Number of participants in which another stone breakage device was used in addition to the study-assigned lithotrite
Time Frame: Intra-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand
Number analyzed (Participants) | 64 | 66 | 71
Participants | 8 | 9 | 5

7. Secondary Outcome: EBL>400mL
Description: Number of participants with an estimated blood loss greater than 400mL
Time Frame: Intra-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand
Number analyzed (Participants) | 64 | 66 | 71
Participants | 4 | 2 | 3

8. Secondary Outcome: RBC Transfusion
Description: Number of participants who required a blood transfusion post-operatively
Time Frame: Post-operatively <24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand
Number analyzed (Participants) | 64 | 66 | 71
Participants | 3 | 2 | 2

9. Secondary Outcome: Length of Stay
Description: Number of days participants were in hospital. Operative day is Day 1.
Time Frame: Post-operatively
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand
Number analyzed (Participants) | 64 | 66 | 71
Days | 1.9 (1.5) | 2.5 (2.1) | 2.6 (2.5)

10. Secondary Outcome: Post-operative Complications
Description: Number of participants who experienced surgery-related post-op complications
Time Frame: Post-operative Days 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand
Number analyzed (Participants) | 64 | 66 | 71
Participants | 10 | 10 | 11

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Stonebreaker | Lithoclast Select | Cyberwand
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/66 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/66 | 0/71
Other Adverse Events (participants affected / at risk) | 18/64 | 19/66 | 16/71
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stonebreaker (N=64) | Lithoclast Select (N=66) | Cyberwand (N=71)
Use of another stone breakage device intraoperatively (Renal and urinary disorders) | 8 | 9 | 5
Post-operative Complications (Surgical and medical procedures) | 10 | 10 | 11 — Number of participants who experienced post-operative complications

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No